CLINICAL TRIAL: NCT06723314
Title: Evaluation of Patient Morbidity and Root Coverage Outcomes of Vestibular Incision Sub Periosteal Tunnel Access Versus Coronally Advanced Flap in Treating Gingival Recession in Esthetic Zone, Randomized Clinical Trial
Brief Title: Evaluation of Patient Morbidity and Root Coverage Outcomes of VISTA Versus CAF in Treating Gingival Recession
Acronym: VISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/2017
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Esthetic Zone
Keywords: recession , gingival recession; connective tissue graft; coronally advanced flap; patient morbidity
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The surgeon performing the surgical technique as well as the patient cannot be blinded because the two surgical procedures are different and recognizable by both the surgeon and the patient after being well informed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Subperiosteal Tunnel Access (Experimental): Vestibular Subperiosteal Tunnel Access
  Interventions: Procedure: Vestibular Subperiosteal Tunnel Access vista
- Coronally Advanced Flap (Active Comparator): Coronally Advanced Flap
  Interventions: Procedure: Vestibular Subperiosteal Tunnel Access vista

INTERVENTIONS:
Procedure: Vestibular Subperiosteal Tunnel Access vista — CAF procedures were performed (Split-Full-Split flap), following the anesthetic agent, the sulcular incision was performed by a full thickness vertical incision till the muccogingival junction• Split thickness releasing incision was made at the flap base with full thickness flap reflection till the muccogingival junction.
  Other Names: coronally advanced flap

SUMMARY:
To evaluate and compare Vestibular Incision Subperiosteal Tunnel Access (VISTA) technique,with connective tissue graft; versus Coronally Advanced Flap (CAF) technique;with connective tissue graft, in treating gingival recession in esthetic zone. Patients and Methods: Thirty patients, with Miller class I or class II gingival recession, were included in the current study, with age range from 18 to 55 years. Defects were treated using either VISTA combined with connective tissue graft technique, or CAF combined with connective tissue technique. Post-operative discomfort was evaluated using the Visual Analog Scale (VAS) to assess patient morbidity. At baseline, 3, 6 and 9 months, clinical parameters were assessed; Probing Depth (PD), Clinical Attachment Level (CAL), Gingival recession Height (GH), Keratinized Tissue Height (KTH), while Complete and Mean Root Coverage (CRC, MRC) were recorded after nine months. Results: The present study revealed that VISTA showed higher significant difference in pain.VISTA also showed a more reduction in PD, CAL, GH as well as KTH than that of CAF with no significant difference between either of the groups.

DETAILED DESCRIPTION:
To evaluate and compare Vestibular Incision Subperiosteal Tunnel Access (VISTA) technique,with connective tissue graft; versus Coronally Advanced Flap (CAF) technique;with connective tissue graft, in treating gingival recession in esthetic zone. Patients and Methods: Thirty patients, with Miller class I or class II gingival recession, were included in the current study, with age range from 18 to 55 years. Defects were treated using either VISTA combined with connective tissue graft technique, or CAF combined with connective tissue technique. Post-operative discomfort was evaluated using the Visual Analog Scale (VAS) to assess patient morbidity. At baseline, 3, 6 and 9 months, clinical parameters were assessed; Probing Depth (PD), Clinical Attachment Level (CAL), Gingival recession Height (GH), Keratinized Tissue Height (KTH), while Complete and Mean Root Coverage (CRC, MRC) were recorded after nine months. Results: The present study revealed that VISTA showed higher significant difference in pain.VISTA also showed a more reduction in PD, CAL, GH as well as KTH than that of CAF with no significant difference between either of the groups. Conclusions: Based on the results of the current study, it can be concluded that both techniques allow improvement in root coverage with no significant differences between them, while VISTA technique showed more pain scores by the VAS than that of CAF technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18- 55 years
* No sexual discrepancy
* Medically free
* Good oral hygeine
* Sound teeth with single (measuring ≥ 2 mm) or Multiple (measuring ≥ 1 mm)
* Class I or II gingival recession defects and adequate amount of keratinized tissue (3mm width).

Exclusion Criteria:

* Patients on anticoagulants, antiplatelets, or glucocorticoids.
* Pregnant females or lactating female patients
* Smoking patients.
* Patients with parafunctional habits.
* Tooth extraction in the surgical sites, active periodontal disease or history of previous surgery in the same area.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Pain Score | 1-10 days
  Visual Analogue Scale to measure pain from (0-10) with 0 (no pain) and 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International Unversity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No